CLINICAL TRIAL: NCT05572918
Title: Translation of a Novel Overactive Bladder 'Fingerprint' Into a Breakthrough Non-invasive Diagnostic Test for Use in a Point of Care Setting
Brief Title: Developing a Simple Test to Diagnose Overactive Bladder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Teesside University (Other)
Collaborators: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, John S. Young, Professor of Translational Healthcare, Teesside University
Other Study IDs: 11043
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Detrusor Overactivity
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mid-stream urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urodynamics aka filling cystometry — Participants will be undergoing a routine diagnostic test to characterise bladder function and volume

SUMMARY:
In order to develop a test to diagnose overactive bladder from urine, it is essential that this test is at least as accurate as the tools that clinicians currently use. As such, this study will compare the performance of the device in development to the performance of existing methods.

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing and able to give informed consent for participation in the study
* The participant has been diagnosed with over-active bladder
* Aged 18 years or above
* Male or Female

Exclusion Criteria:

* The participant is unwilling to give informed consent for participation in the study
* The participant is unable to represent their own interests or is particularly susceptible to coercion (i.e. is deemed as vulnerable)
* The participant has been diagnosed with neurologic disease (stroke, MS, Parkinson's disease, spinal cord injury); history of uterine, cervical, vaginal or urethral cancer; history of cyclophosphamide use or any type of chemical cystitis; history of benign or malignant bladder tumours; has had Botulinum injections, neuromodulation or augmentation cystoplasty
* Aged 17 years or younger.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients with urinary symptoms referred to Consultant Urological Surgeon Ms Mehwash Nadeem at the James Cook Hospital, Middlesbrough or the Friarage Hospital, Northallerton, to undergo a diagnostic test to characterise bladder function and volume.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of accuracy of a diagnostic test for overactive bladder | December 2022 - November 2023
  A prototype lateral flow immunoassay dipstick to detect specific urinary biomarkers for OAB, based on specific urinary biomarkers and with a dynamic range and sensitivity required for accurate OAB diagnosis.

IPD SHARING:
Plan to Share IPD: No